CLINICAL TRIAL: NCT00550043
Title: A Double-blind, Placebo-controlled Study Exploring the Safety, Tolerability and Efficacy of a 4 Week Course of INCB018424 in Subjects With Active Rheumatoid Arthritis
Brief Title: A Study Exploring the Safety, Tolerability and Efficacy of a 4 Week Course of INCB018424 in Subjects With Active Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: INCB 18424-231
Record Dates: First submitted 2007-10-24; First posted 2007-10-26 (Estimated); Results first posted 2015-03-23 (Estimated); Last update posted 2015-03-23 (Estimated); Status verified 2015-03

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — ruxolitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Cohort 1: Treatment Group A (Experimental): INCB018424 15 mg twice daily (BID) or matching placebo
  Interventions: Drug: INCB018424
- Cohort 2: Treatment Group B (Experimental): INCB018424 5 mg BID or matching placebo
  Interventions: Drug: INCB018424
- Cohort 2: Treatment Group C (Experimental): INCB018424 25 mg BID or matching placebo
  Interventions: Drug: INCB018424
- Cohort 2: Treatment Group D (Experimental): INCB018424 50 mg once daily (QD) or matching placebo
  Interventions: Drug: INCB018424
- Placebo (Placebo Comparator): Matching placebo, oral
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: INCB018424
  Arms: Cohort 1: Treatment Group A; Cohort 2: Treatment Group B; Cohort 2: Treatment Group C; Cohort 2: Treatment Group D
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to understand the safety and tolerability of INCB018424 in patients with rheumatoid arthritis

ELIGIBILITY:
Inclusion Criteria:

1. Established diagnosis of rheumatoid arthritis
2. Patients receiving methotrexate must be treated with for at least 6 months and receiving a stable weekly dose between 10 and 25 mg for at least 8 consecutive weeks prior to study entry.

Exclusion Criteria:

1. Patients who have taken the following drugs within the timeframe below:

   * Leflunomide, infliximab, etanercept, adalimumab, abatacept, or other biological therapies (except rituximab) - Within 12 weeks prior to the first dose of study medication;
   * Rituximab - Within 12 months prior to the first dose of study medication;
   * Disease-modifying anti-rheumatic drugs (DMARDs) or other anti-rheumatic therapies not specified above including but not limited to: gold, penicillamine, dapsone, azathioprine, 6-mercaptopurine, chlorambucil, cyclophosphamide, cyclosporin, mycophenolate mofetil - Within 12 weeks prior to the first dose of study medication;
2. Treatment with any investigational medication within 12 weeks prior to the first dose of study medication.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2007-10; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Monica Luchi, MD, Study Director — Incyte Corporation
Locations (15):
- United States (12):
  - Huntsville, Alabama
  - Upland, California
  - Gainesville, Florida
  - Palm Harbor, Florida
  - Kalispell, Montana
  - Hickory, North Carolina
  - Mayfield Village,, Ohio
  - Middleburg Heights, Ohio
  - Perrysburg, Ohio
  - Pittsburgh, Pennsylvania
  - Hixson, Tennessee
  - Memphis, Tennessee
- Poland (3):
  - Elblag
  - Gmina Końskie
  - Warsaw

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: Treatment Group A: INCB018424 15 mg BID
- Cohort 2: Treatment Group B: INCB018424 5 mg BID
- Cohort 2: Treatment Group C: INCB018424 25 mg BID
- Cohort 2: Treatment Group D: INCB018424 50 mg QD
Period: Overall Study
Arm/Group | Placebo | Cohort 1: Treatment Group A | Cohort 2: Treatment Group B | Cohort 2: Treatment Group C | Cohort 2: Treatment Group D
Started | 9 | 12 | 9 | 10 | 10
Completed | 9 | 9 | 8 | 8 | 9
Not Completed | 0 | 3 | 1 | 2 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 1
Not completed — Subject Withdrew Consent | 0 | 2 | 1 | 0 | 0
Not completed — Other Reasons- Unspecified | 0 | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Cohort 1: Treatment Group A | Cohort 2: Treatment Group B | Cohort 2: Treatment Group C | Cohort 2: Treatment Group D | Total
Number analyzed (Participants) | 9 | 12 | 9 | 10 | 10 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.2 (12.04) | 56.9 (8.44) | 49.6 (10.69) | 57.5 (11.29) | 54.5 (14.14) | 54.9 (11.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 7 | 7 | 8 | 38
  Male | 1 | 4 | 2 | 3 | 2 | 12

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Subjects Achieving American College of Rheumatology (ACR) 20 Improvement
Description: The ACR 20 is defined as ≥ 20% improvement in tender joint count plus ≥ 20% improvement in swollen joint count plus ≥ 20% improvement in 3 of the following 5 criteria: subject's assessment of pain, Subject's global assessment of disease activity (PGA), Physician's global assessment of disease activity (PHGA), subject's self-assessed disability Health Assessment Questionnaire (HAQ), and Erythrocyte sedimentation rate (ESR) or C-reactive protein (CRP), whichever shows the greatest change.
Time Frame: Day 28
Population: modified intent-to-treat (mITT) Population: subjects enrolled, took 1 dose of study drug, had predose and at least 1 post baseline Rheumatoid arthritis (RA) assessments. Subjects discontinuing before the last scheduled efficacy evaluation had data imputed for time points after discontinuation; they had their last observation carried forward (LOCF).
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Cohort 1: Treatment Group A | Cohort 2: Treatment Group B | Cohort 2: Treatment Group C | Cohort 2: Treatment Group D
Number analyzed (Participants) | 9 | 12 | 9 | 10 | 10
Percentage of participants
  No Response | 66.7 | 16.7 | 66.7 | 40.0 | 40.0
  Response | 33.3 | 83.3 | 33.3 | 60.0 | 60.0

2. Secondary Outcome: The Percentage of Subjects Achieving ACR 50 Improvement
Description: The ACR 50 is defined as ≥ 50% improvement in tender joint count plus ≥ 50% improvement in swollen joint count plus ≥50% improvement in 3 of the following 5 criteria: subject's assessment of pain, PGA, PHGA, subject's self-assessed disability HAQ, and ESR or CRP, whichever shows the greatest change.
Time Frame: Day 28
Population: mITT Population: subjects who were enrolled, took at least 1 dose of study drug, and had predose and at least 1 post baseline Rheumatoid arthritis (RA) assessments. Subjects who discontinued before the last scheduled efficacy evaluation had data imputed for time points after discontinuation; they had their last observation carried forward (LOCF).
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Cohort 1: Treatment Group A | Cohort 2: Treatment Group B | Cohort 2: Treatment Group C | Cohort 2: Treatment Group D
Number analyzed (Participants) | 9 | 12 | 9 | 10 | 10
Percentage of participants
  No Response | 88.9 | 50.0 | 88.9 | 60.0 | 50.0
  Response | 11.1 | 50.0 | 11.1 | 40.0 | 50.0

3. Secondary Outcome: The Percentage of Subjects Achieving ACR 70 Improvement
Description: The ACR 70 is defined as ≥ 70% improvement in tender joint count plus
  ≥ 70% improvement in swollen joint count plus ≥ 70% improvement in 3 of the following 5 criteria: subject's assessment of pain, PGA, PHGA, subject's self-assessed disability HAQ, and ESR or CRP, whichever shows the greatest change.
Time Frame: Day 28
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Cohort 1: Treatment Group A | Cohort 2: Treatment Group B | Cohort 2: Treatment Group C | Cohort 2: Treatment Group D
Number analyzed (Participants) | 9 | 12 | 9 | 10 | 10
Percentage of participants
  No response | 100.0 | 75.0 | 100.0 | 70.0 | 70.0
  Response | 0.0 | 25.0 | 0.0 | 30.0 | 30.0

4. Secondary Outcome: Change From Baseline in Disease Activity Score 28 (DAS 28) ESR Score
Description: Calculation of the disease activity score 28 (DAS 28) score was based on the tender joint count, plus swollen joint count, plus PGA, plus Erythrocyte sedimentation rate (ESR). The DAS28-ESR is expressed as units on a scale with the minimum score=0 (best) to maximum score=10 (worst). Remission was defined as DAS28-ESR <2.6. The mean change from baseline (which represent decreases in the DAS 28 ESR scores) are shown as positive numbers in these analyses.
Time Frame: Baseline, Day 28
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Cohort 1: Treatment Group A | Cohort 2: Treatment Group B | Cohort 2: Treatment Group C | Cohort 2: Treatment Group D
Number analyzed (Participants) | 9 | 12 | 9 | 10 | 10
Units on a scale | 1.32 (0.845) | 2.72 (1.250) | 1.09 (1.107) | 2.53 (1.454) | 2.88 (1.225)

5. Secondary Outcome: Change From Baseline in Disease Activity Score 28 (DAS 28) CRP Score
Description: Calculation of the disease activity score 28 (DAS 28) score was based on the tender joint count, plus swollen joint count, plus PGA, plus C-reactive protein (CRP). A higher score indicated more disease activity. The mean change from baseline (which represent decreases in the DAS 28 CRP scores) are shown as positive numbers in these analyses. The DAS28 provides a score on a scale from 0 to 10 indicating the current activity of the rheumatoid arthritis (>5.1=high disease activity; <3.2=low disease activity; <2.6=remission).
Time Frame: Baseline, Day 28
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Cohort 1: Treatment Group A | Cohort 2: Treatment Group B | Cohort 2: Treatment Group C | Cohort 2: Treatment Group D
Number analyzed (Participants) | 9 | 12 | 9 | 10 | 10
Units on a scale | 1.14 (0.907) | 2.27 (1.177) | 0.92 (0.985) | 2.33 (1.840) | 2.64 (1.275)

6. Secondary Outcome: Percentage of Subjects Who Achieved DAS 28 ESR Low Disease
Description: Subjects who achieved low disease activity based on the DAS 28 ESR (score <3.2). Subjects who achieved low disease activity were classified as responders in this analysis.
Time Frame: Day 28
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Cohort 1: Treatment Group A | Cohort 2: Treatment Group B | Cohort 2: Treatment Group C | Cohort 2: Treatment Group D
Number analyzed (Participants) | 9 | 12 | 9 | 10 | 10
Percentage of participants
  Non-responders | 100.0 | 50.0 | 100.0 | 90.0 | 60.0
  Responders | 0.0 | 50.0 | 0.0 | 10.0 | 40.0

7. Secondary Outcome: Percentage of Subjects Who Achieved DAS 28 CRP Low Disease
Description: Subjects who achieved low disease activity based on the DAS 28 CRP (score <3.2). Subjects who achieved low disease activity were classified as responders in this analysis.
Time Frame: Day 28
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Cohort 1: Treatment Group A | Cohort 2: Treatment Group B | Cohort 2: Treatment Group C | Cohort 2: Treatment Group D
Number analyzed (Participants) | 9 | 12 | 9 | 10 | 10
Percentage of participants
  Non-responders | 100.0 | 50.0 | 100.0 | 70.0 | 50.0
  Responders | 0.0 | 50.0 | 0.0 | 30.0 | 50.0

8. Secondary Outcome: Percentage of Subjects Who Achieved DAS 28 ESR Inactive Disease
Description: Subjects who achieved inactive disease based on the DAS 28 ESR (score <2.6). Subjects who achieved low disease activity were classified as responders in this analysis.
Time Frame: Day 28
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Cohort 1: Treatment Group A | Cohort 2: Treatment Group B | Cohort 2: Treatment Group C | Cohort 2: Treatment Group D
Number analyzed (Participants) | 9 | 12 | 9 | 10 | 10
Percentage of participants
  Non-responders | 100.0 | 75.0 | 100.0 | 100.0 | 90.0
  Responders | 0.0 | 25.0 | 0.0 | 0.0 | 10.0

9. Secondary Outcome: Percentage of Subjects Who Achieved DAS 28 CRP Inactive Disease
Description: Subjects who achieved inactive disease based on DAS 28 CRP (score <2.6). Subjects who achieved low disease activity were classified as responders in this analysis.
Time Frame: Day 28
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Cohort 1: Treatment Group A | Cohort 2: Treatment Group B | Cohort 2: Treatment Group C | Cohort 2: Treatment Group D
Number analyzed (Participants) | 9 | 12 | 9 | 10 | 10
Percentage of participants
  Non-responders | 100.0 | 75.0 | 100.0 | 90.0 | 70.0
  Responders | 0.0 | 25.0 | 0.0 | 10.0 | 30.0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time the subject ingested the first dose of study drug up to 28 days after the last dose of study drug was administered.
Description: Treatment-Emergent Adverse Events are those that either newly occurred after the first study drug dosing, or worsened from baseline
Arm/Group | Placebo | Cohort 1: Treatment Group A | Cohort 2: Treatment Group B | Cohort 2: Treatment Group C | Cohort 2: Treatment Group D
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/12 | 0/9 | 0/10 | 1/10
Other Adverse Events (participants affected / at risk) | 5/9 | 6/12 | 2/9 | 6/10 | 7/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=9) | Cohort 1: Treatment Group A (N=12) | Cohort 2: Treatment Group B (N=9) | Cohort 2: Treatment Group C (N=10) | Cohort 2: Treatment Group D (N=10)
Congestive cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 — Congestive cardiac failure and Interstitial lung disease were reported in the same subject 3 weeks after the last dose of study medication and resolved 2 weeks later.
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 — Congestive cardiac failure and Interstitial lung disease were reported in the same subject 3 weeks after the last dose of study medication and resolved 2 weeks later.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=9) | Cohort 1: Treatment Group A (N=12) | Cohort 2: Treatment Group B (N=9) | Cohort 2: Treatment Group C (N=10) | Cohort 2: Treatment Group D (N=10)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Ocular hyperaemia (Eye disorders) | 1 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Breath odour (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 2 | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0
Blood cholesterol increased (Investigations) | 0 | 0 | 0 | 0 | 1
Haematocrit decreased (Investigations) | 0 | 0 | 0 | 2 | 0
Haemoglobin decreased (Investigations) | 1 | 0 | 0 | 2 | 1
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 1 | 0
Mean cell haemoglobin concentration decreased (Investigations) | 0 | 0 | 0 | 1 | 0
Mean cell volume increased (Investigations) | 0 | 0 | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 1 | 0
Occult blood positive (Investigations) | 0 | 0 | 0 | 1 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 1
Red blood cell count decreased (Investigations) | 0 | 0 | 0 | 1 | 0
Red cell distribution width increased (Investigations) | 0 | 0 | 0 | 1 | 0
Reticulocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 1
Reticulocyte count increased (Investigations) | 0 | 0 | 0 | 1 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Renal colic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Mass excision (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following the first publication, the Institution and/or Principal Investigator may publish data or results from the Study, provided, however, that the Institution and/or Principal Investigator submits the proposed publication to the Sponsor for review at least sixty (60) days prior to the date of the proposed publication. Sponsor may remove from the proposed publication any information that is considered confidential and/or proprietary other than Study data and results.